CLINICAL TRIAL: NCT01663090
Title: Ferumoxytol-Enhanced Magnetic Resonance Imaging (MRI) in Pediatric and Adult Patients With Malignant Sarcoma: A Two-part Pilot Study for Safety and Efficacy in the Pediatric and Adult Populations
Brief Title: Ferumoxytol-Enhanced MRI in Adult/Pedi Sarcomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to accrue.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Allison O'Neill, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-254
Record Dates: First submitted 2012-07-28; First posted 2012-08-13 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: Newly diagnosed
MeSH Terms: conditions — Sarcoma | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nanoparticle enhanced MRI (Experimental)
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol

SUMMARY:
This research study is a pilot study to evaluate a new contrast agent, ferumoxytol, for the purpose of imaging lymph node metastases in patients with soft tissue sarcoma. This contrast agent is an investigational drug. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved ferumoxytol for this use. This drug has been used to image adults with other forms of cancer, however, it has only been used to image a small number of pediatric patients. Ferumoxytol has never been used to image sarcoma.

DETAILED DESCRIPTION:
Before the research starts you will undergo some screening procedures to confirm that you are eligible to participate in the study. These include a medical history, blood tests and an electrocardiogram.

After we confirm taht you are eligible for this study you will undergo the following. We estimate that you will be on the study for approximately two to three weeks.

Baseline MRI of the tumor site and draining lymph nodes: Whether you are on the study or not you will have a baseline MRI which involves the use of a standard contrast agent called gadolinium. This imaging test is considered the standard of care and is the method by which doctors determine tumor location and spread. This MRI is NOT part of the study.

Ferumoxytol Infusion: You will receive this study drug the same day as your baseline MRI; if you already had your baseline MRI, this medication can be given intravenously (i.e. directly into the vein) at your next clinical visit. It can likewise be given through a central line. You will be observed during the infusion and 30 minutes after the infusion to ensure that you do not have an allergic or adverse reaction to the medication.

Repeat MRI of the tumor site and draining lymph nodes: Three to five days after receiving ferumoxytol, you will undergo a repeat MRI. You will not require any additional contrast prior to this imaging study. This MRI is part of the study.

Lymph Node Biopsy: You will be undergoing a lymph node biopsy whether or not you are on the study. This will occur approximately a week after your study MRI. This is a surgical procedure that involves removing one or a few lymph nodes in the region of your tumor and studying them under a microscope to determine whether they contain signs of microscopic cancer spread. Your surgeon will explain this procedure to you in more detail.

We anticipate that your clinic visit for ferumoxytol will take approximately an hour. MRI tests, on average, likewise take approximately an hour to complete.

After you have completed the study MRI and lymph node biopsy, you will require one additional blood test to measure blood iron levels. We measure iron levels because ferumoxytol is comprised of an iron core. This iron is similar to that in oral iron supplements and can cause your blood iron levels to temporarily increase. Because we are trying to determine whether this contrast agent will be useful, you will not receive teh results to the study MRI. If however, lymph nodes are found to be positive for disease, your treatment plan may change to address this.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of soft tissue sarcoma, who will undergo lymph node biopsy
* Able to tolerate MRI scan without sedation/anesthesia
* Greater than or equal to 12 years of age

Exclusion Criteria:

* Previous therapy other than biopsy or surgical resection of the primary tumor
* Pregnant or breastfeeding
* Receipt of other iron-oxide based nanoparticle therapy within 4 weeks of scans
* History of allergic reaction to compounds of similar composition to ferumoxytol
* Known diagnosis of hemochromatosis, mitochondrial disorder or iron overload
* Invasive bacterial infection
* Known history of contrast sensitivity
* Braces or metal heart valve that may interfere with MRI, surgical clips, a pacemaker, piercings that cannot be removed, or any other indwelling metal device that might interfere with MRI

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and sensitivity of nanoparticle-enhanced MRI | 4 years
  To determine the feasibility and evaluate the sensitivity of using nanoparticle-enhanced MRI in detecting lymph node metastases in pediatric and adult soft tissue sarcoma patients with clinically palpable or radiographically concerning lymph nodes, whereby the minimum acceptable sensitivity was selected based on a histologic gold standard
Sensitivity of nanoparticle-enhanced MRI in occult lymph node metastases | 4 years
  To evaluate the sensitivity of nanoparticle-enhanced MRI in detecting occult lymph node metastases in pediatric and adult patients with soft tissue sarcoma, whereby the minimum acceptable sensitivity was selected based on a histologic gold standard

SECONDARY OUTCOMES:
Safety of ferumoxytol in pediatric patients | 4 years
  The safety of ferumoxytol in pediatric patients will be assessed by the proportion of patients who experience at least one dose limiting toxicity (DLT). DLT refers to toxicities experienced after the start of the drug infusion; they are based on the Common Terminology Criteria for Adverse Events version 4.0.
Sensitivity of conventional MRI vs. nanoparticle enhanced MRI | 4 years
  To evaluate the sensitivity of conventional MRI in detecting the presence of lymph node abnormalities in pediatric and adult patients with soft tissue sarcoma, and to compare this to the sensitivity of nanoparticle-enhanced MRI. The sensitivity of nanoparticle-enhanced MRI will be descriptively compared to the sensitivity of conventional MRI, where in each case the histological confirmation of lymph node involvement is the "standard of truth." For conventional MRI, sensitivity will be measured by the number of patients in whom at least one lymph node abnormality was detected by conventional MRI, as determined by the primary radiologist, divided by the total number of evaluable patients.
Compare inter-reader variability in the interpretation of nanoparticle MRI scans | 4 years
  To determine inter-reader variability in the interpretation of nanoparticle MRI scans by two independent radiologists. The comparison will be made between each central review radiologist's assessment of whether or not a given patient has a positive lymph node.
Retrospective central pathology review | 4 years
  To perform a retrospective central pathology review to determine inter-pathologist interpretation of positive lymph nodes. This too will be done through comparison of each central review pathologist's assessment of whether or not a given patient has a positive lymph node.

CONTACTS AND LOCATIONS:
Overall Officials: Allison O'Neill, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts